CLINICAL TRIAL: NCT05647447
Title: Pilot of Osanetant to Reduce Severity of Hot Flashes in Men With Adenocarcinoma of the Prostate (POSH-MAP)
Brief Title: Pilot of Osanetant to Reduce Severity of Hot Flashes in Men With Adenocarcinoma of the Prostate
Acronym: POSH-MAP
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Development of the drug program has been discontinued
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00148766
Record Dates: First submitted 2022-11-01; First posted 2022-12-12 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — SR 142801

STUDY DESIGN:
Intervention Model Description: Single-arm pilot
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pilot Trial: Osanetant 28 Days (Experimental): Osanetant 200 mg orally, twice per day for 28 days.
  Interventions: Drug: Osanetant

INTERVENTIONS:
Drug: Osanetant — Osanetant 200 mg orally, twice per day

SUMMARY:
To evaluate the preliminary efficacy of in reducing the frequency and severity of hot flashes in men on androgen deprivation therapy (ADT).

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent
* Males ≥ 18 years
* Histologic diagnosis of prostate cancer (PCa)
* Undergoing active treatment with ADT within ≥ 30 days prior to randomization
* Using either an gonadotropin releasing hormone (GNRH) agonist with a planned duration covering the 8 weeks of the study or are status post bilateral orchiectomy,
* Have a castrate level of testosterone (≤ 50 ng/dL) at enrollment
* Have moderate-to-severe hot flashes defined as

  * Seven (7) or more hot flashes per day
  * Total hot flash severity (HFS: total number of hot flashes for 1 week multiplied by the average severity/week) ≥ 100
* Adequate organ function, defined as follows: Result Date

  * Leukocytes > 1.5K/UL
  * Absolute Neutrophil Count (ANC) >1.5K/UL NOTE: Patients with established diagnosis of benign neutropenia are eligible to participate with ANC between 1000-1500 if in the opinion of treating physician the trial treatment does not pose excessive risk of infection to the patient.
  * Platelets >100K/UL
  * Hemoglobin ≥ 9 g/dL
  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault equation
  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault equation
  * Total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ 1 x ULN
  * Aspartate aminotransferase and alanine aminotransferase ≤ 1.5 x ULN
* Women of child-bearing potential and men with partners of childbearing potential must agree to practice sexual abstinence or to use the forms of contraception listed in Child-Bearing Potential/Pregnancy section for the duration of study participation and for 30 days following completion of therapy.

Exclusion Criteria:

* Concurrent invasive malignancy or invasive malignancy within 2 years except for chronic lymphocytic leukemia/small lymphocytic lymphoma on surveillance, suspected or proven clinical stage 1 (cT1) renal cell carcinoma on active surveillance, or the following malignancies treated with curative intent via surgical resection: carcinoma in situ of the cervix, ductal carcinoma in situ of the breast, low-grade non-muscle-invasive urothelial carcinoma, non-melanoma skin cancer.
* Simultaneously enrolled in any therapeutic clinical trial
* Current or anticipating use of other pharmacologic anti-neoplastic (including hormonal), or investigational agents while participating in this study. Concurrent treatment with radiotherapy is permitted.
* Diagnosed with a psychiatric illness or is in a social situation that would limit compliance with study requirements
* Has a known allergic reaction to any excipient contained in the study drug formulation
* Active Grade 3 (per the NCI CTCAE, Version 5.0) or higher viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study treatment.
* Participants using the following medications within 2 weeks prior to first dosing (or within 5 times the half-life of that medication, whichever is longer) will be excluded from the study:

  * Inhibitors of CYP3A4 (including but not limited to macrolide antibiotics, HIV protease inhibitor, azole antifungal drugs, cyclosporine, calcium channel inhibitor, cimetidine)
  * Inducers of CYP3A4 (including but not limited to rifampicin, carbamazepine, efavirenz, bosentan, modafinil, St. John's Wort), Medications with narrow therapeutic index that are metabolized CYP3A4 and/or CYP2D6 are not allowed from screening until up to 5 half-lives after last dose of Osanetant is administered.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the preliminary efficacy of in reducing the frequency and severity of vasomotor symptoms (VMS) in men on androgen deprivation therapy (ADT). | 28 days
  Efficacy will be assessed using a composite outcome of median weekly hot flash frequency and severity at week 4 compared to baseline.

SECONDARY OUTCOMES:
To evaluate the effect of Osanetant on follicle stimulating hormone for men with prostate cancer on ADT. | 28 days
  Levels of follicle stimulating hormone (FSH) will be measured at week 4 will be compared to baseline.
To evaluate the effect of Osanetant on luteinizing hormone for men with prostate cancer on ADT. | 28 days
  luteinizing hormone (LH) will be measured at week 4 will be compared to baseline.
To evaluate the effect of Osanetant on testosterone for men with prostate cancer on ADT. | 28 days
  testosterone will be measured at week 4 will be compared to baseline.
To evaluate the effect of Osanetant on estradiol for men with prostate cancer on ADT. | 28 days
  estradiol will be measured at week 4 will be compared to baseline. with prostate cancer on ADT
Functional Assessment of Cancer Therapy-Prostate (FACT-P) | 28 days
  To evaluate the impact of Osanetant on global quality of life with Functional Assessment of Cancer Therapy-Prostate (FACT-P)
EuroQOL 5-dimension | 28 days
  To evaluate the impact of Osanetant on global quality of life with a visual analog scale from EuroQOL 5-dimension, 5-level (EQ-5D-5L). The EQ-5D-5L visual analog scale is 0-100 with higher numbers being better.
Patient Health Questionnaire-9 question (PHQ-9). | 28 days
  To evaluate the impact of Osanetant on depressive symptoms on Patient Health Questionnaire-9 question (PHQ-9).
General Anxiety Disorder-7 question (GAD-7) | 28 days
  To evaluate the impact of Osanetant on anxiety symptoms on General Anxiety Disorder-7 question (GAD-7).
Hot Flash Related Daily Interference Scale (HFRDIS). | 28 days
  To evaluate the impact of Osanetant on hot flash interference using the Hot Flash Related Daily Interference Scale (HFRDIS). The hot flash daily interference scale has a minimum of 0 and a max of 100, with higher scores indicating more interference (which is worse).

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas, United States